CLINICAL TRIAL: NCT05431790
Title: Absorbable Interface Screw Clinical Trial - PUTH & NANTON
Brief Title: Absorbable Interface Screw Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00006761-D2022055
Record Dates: First submitted 2022-05-31; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-05

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Anterior cruciate ligament; absorbable interface screws
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Random assignment of patients with anterior cruciate ligament reconstruction (The test group uses the test product; the control group uses the marketed product)Blind the subjects.
Who Masked: Participant
Masking Description: Blind the participant (Due to the particularity of implanted devices, blindness needs to be maintained as far as possible until the subject is automatically unblinded)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Absorbable screw (Natong Biotechnology (Beijing) Co., Ltd.) (Experimental): Anterior cruciate ligament reconstruction uses absorbable interface screws manufactured by Natong Biotechnology.
  Interventions: Device: Absorbable interface screws manufactured by Natong Biotechnology
- Absorbable screw (Inion Oy, INION, Finland) (Active Comparator): Anterior cruciate ligament reconstruction uses absorbable interface screws manufactured by INION.
  Interventions: Device: Absorbable interface screws manufactured by INION.

INTERVENTIONS:
Device: Absorbable interface screws manufactured by Natong Biotechnology — Anterior cruciate ligament reconstruction uses absorbable interface screws manufactured by Natong Biotechnology.
  Arms: Absorbable screw (Natong Biotechnology (Beijing) Co., Ltd.)
Device: Absorbable interface screws manufactured by INION. — Reconstruction of anterior cruciate ligament using Inion Oy absorbable interface scews from INION, Finland
  Arms: Absorbable screw (Inion Oy, INION, Finland)

SUMMARY:
Validation of the safety and efficacy of absorbable interface screws for clinical use

DETAILED DESCRIPTION:
Interface screws are divided into metal screws and absorbable screws. Since metal screws cut tendon grafts, absorbable interface screws are now mostly selected. At present, the materials of absorbable screws are mainly polylactic acid and polyglycolide. The test product is composed of two kinds of polylactic acid and bioactive glass fiber, which can reduce the adverse stimulation to the surrounding bone, promote the absorption of the screw and the bone grow into.Estimated enrollment for 4 months, follow-up for 14 months, a total of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* ① Before surgery, subjects or guardians are willing and able to sign the informed consent;

  * Patients aged 18 to 80 (including 18 and 80 years old), regardless of gender;

    * Patients who meet the diagnostic criteria for anterior cruciate ligament rupture of the knee joint and have no contraindications to implantation;

      * The patient's bones are mature;

        * Good compliance, willing and able to conduct follow-up observation as required.

Exclusion Criteria:

* ① Subjects who have participated in other clinical studies of drugs, biological agents or medical devices before being selected and did not reach the primary study endpoint;

  * The patient is known to have a history of allergy to one or more implanted materials;

    * Those who are physically weak or cannot tolerate surgery due to other diseases of the body;

      * Active infection in the knee joint or other parts of the body; ⑤ Those with other ligament injury and/or meniscus injury in the affected knee joint; ⑥ Those who need to perform simultaneous meniscus repair and other surgeries on the ipsilateral knee joint; ⑦ Obese BMI>35;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Lysholm score | Asked as baseline data before surgery.
  An instrument used to assess the results of rehabilitation from knee injuries, especially those requiring ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION. It measures recovery of knee joint function based on ACTIVITIES OF DAILY LIVING.
  Year introduced: 2015 Patients will be asked to fill out the Lysholm score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Lysholm score | At 6 months after surgery.
  An instrument used to assess the results of rehabilitation from knee injuries, especially those requiring ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION. It measures recovery of knee joint function based on ACTIVITIES OF DAILY LIVING.
  Year introduced: 2015 Patients will be asked to fill out the Lysholm score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Lysholm score | At 9 months after surgery.
  An instrument used to assess the results of rehabilitation from knee injuries, especially those requiring ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION. It measures recovery of knee joint function based on ACTIVITIES OF DAILY LIVING.
  Year introduced: 2015 Patients will be asked to fill out the Lysholm score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Lysholm score | At 14 months after surgery.
  An instrument used to assess the results of rehabilitation from knee injuries, especially those requiring ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION. It measures recovery of knee joint function based on ACTIVITIES OF DAILY LIVING.
  Year introduced: 2015 Patients will be asked to fill out the Lysholm score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
The upper, middle and lower diameters of the tibial bone tunnel | Preoperatively, 6 months postoperatively, 9 months postoperatively, and 14 months postoperatively.
  The tunnel widening of the experimental group was measured compared with that of the control group.
Relative tibial anterior displacement | Preoperatively, 6 months postoperatively, 9 months postoperatively, and 14 months postoperatively.
  To compare whether the absorbable interface screws in the experimental group can effectively limit the anterior displacement of the tibia relative to the femur.
Range of motion (ROM) | Preoperatively.
  Assessing active and passive flexion-extension angles after anterior cruciate ligament surgery
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form 2000. | Asked as baseline data before surgery.
  Currently, there are internationally recognized scales with reliability, validity and sensitivity for the assessment of anterior cruciate ligament injury and rupture. Subjective and objective symptoms of the knee joint were comprehensively assessed.
Tegner score | Asked as baseline data before surgery.
  Patients will be asked to fill out the Tegner score to document the functional status. The minimum is 0 and the maximum value is 10. Higher scores mean a better outcome.
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form 2000 | At 6 months after surgery.
  Currently, there are internationally recognized scales with reliability, validity and sensitivity for the assessment of anterior cruciate ligament injury and rupture. Subjective and objective symptoms of the knee joint were comprehensively assessed.
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form 2000 | At 9 months after surgery.
  Currently, there are internationally recognized scales with reliability, validity and sensitivity for the assessment of anterior cruciate ligament injury and rupture. Subjective and objective symptoms of the knee joint were comprehensively assessed.
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form 2000 | At 14 months after surgery.
  Currently, there are internationally recognized scales with reliability, validity and sensitivity for the assessment of anterior cruciate ligament injury and rupture. Subjective and objective symptoms of the knee joint were comprehensively assessed.
Tegner score | At 6 months after surgery.
  Patients will be asked to fill out the Tegner score to document the functional status. The minimum is 0 and the maximum value is 10. Higher scores mean a better outcome.
Tegner score | At 9 months after surgery.
  Patients will be asked to fill out the Tegner score to document the functional status. The minimum is 0 and the maximum value is 10. Higher scores mean a better outcome.
Tegner score | At 14 months after surgery.
  Patients will be asked to fill out the Tegner score to document the functional status. The minimum is 0 and the maximum value is 10. Higher scores mean a better outcome.
Relative tibial anterior displacement | At 6 months postoperatively.
  To compare whether the absorbable interface screws in the experimental group
Relative tibial anterior displacement | At 9 months postoperatively.
  To compare whether the absorbable interface screws in the experimental group
Relative tibial anterior displacement | At 14 months postoperatively.
  To compare whether the absorbable interface screws in the experimental group
Range of motion (ROM) | At 6 months postoperatively.
  Assessing active and passive flexion-extension angles after anterior cruciate ligament surgery
Range of motion (ROM) | At 9 months postoperatively.
  Assessing active and passive flexion-extension angles after anterior cruciate ligament surgery
Range of motion (ROM) | At 14 months postoperatively.
  Assessing active and passive flexion-extension angles after anterior cruciate ligament surgery